CLINICAL TRIAL: NCT04341155
Title: Adjunctive Dexamethasone for Cerebral Toxoplasmosis: a Double-blinded Randomized Controlled Trial
Brief Title: Dexamethasone for Cerebral Toxoplasmosis
Acronym: De-Tox
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TX-202003.01
Record Dates: First submitted 2020-03-31; First posted 2020-04-10 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Toxoplasmosis, Cerebral
MeSH Terms: conditions — Toxoplasmosis, Cerebral | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Active Comparator): Sixty nine patients will be administered randomly dexamethasone 20 mg IV for 7 days.
  Along with study drug or placebo, patients will receive standard anti toxoplasmosis (Oral pyrimethamine 150 or 200 mg (according to body weight) for three days continued by 50 or 75mg (according to body weight) per day or oral cotrimoxazole 2 x 1920 mg; oral clindamycin 600mg q.i.d) in accordance to national neurologist association guidelines.
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Sixty nine patients will be administered randomly Normal Saline 0,9% IV (4 cc) for 7 days.
  Along with study drug or placebo, patients will receive standard anti toxoplasmosis (Oral pyrimethamine 150 or 200 mg (according to body weight) for three days continued by 50 or 75mg (according to body weight) per day or oral cotrimoxazole 2 x 1920 mg; oral clindamycin 600mg q.i.d) in accordance to national neurologist association guidelines.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Patients in experimental arms will receive i.v. dexamethasone 20 mg (4 ampules = 20mL) for 7 days
  Other Names: Dexamethasone - Phapros
  Arms: Dexamethasone
Drug: Placebo — Patients in placebo arms will receive 20 mL normal saline intravenously for 7 days
  Other Names: Normal Saline 0,9% - B Braun
  Arms: Placebo

SUMMARY:
Toxoplasma gondii infects over one third of the global human population. Cerebral toxoplasmosis is the most common opportunistic infection in HIV patients resulting in up to 50% of mortality with proper treatment and 80% without it. The fatality mainly due to the brain edema resulted from the mass effect lesion. In addition of anti toxoplasmosis given, adjunctive therapy such as steroid is recommended in order to reduce brain edema, but the dose and duration of administration in cerebral toxoplasmosis has not been evaluated in a clinical trial. Adjunctive therapy given in cerebral toxoplasmosis patients still remains unclear. Moreover, its safety in immunodeficiency cases is still debatable.

DETAILED DESCRIPTION:
Steroid produces a raising expression of anti inflammation genes (NF-κB, IκB-α and antagonist receptor IL-1) and inhibits pro inflammation cytokines ( TNF-α and IL-1β). It also works as anti edema by correcting the disrupted blood brain barrier during infection process. Dexamethasone is considered to be chosen in this clinical trial due to the long half life among steroids, the strongest glucocorticoid effect comparing other steroids, and easily prepared and used on daily practice.

There are limited data from using adjunctive steroid for treatment of HIV-associated with cerebral toxoplasmosis. Previous study in France published in 2012 showed steroid did not give any significant improvement for patients' neurological outcome and did not worsen patients' condition such as getting nosocomial infection. Meanwhile comparing previous study by Arens et. al in 2007, there was an increasing mortality rate on adjunctive steroid used in cerebral toxoplasmosis patients.

As result of limited data, our trial is looked forward to answer about the efficacy of dexamethasone treatment in reducing mortality rate of cerebral toxoplasmosis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or above.
2. Clinical signs and symptoms compatible to cerebral toxoplasmosis
3. Serology HIV positive
4. Immunoglobulin G anti-toxoplasma titre is positive
5. One or more mass lesions on the neuroradiological finding
6. None or less than 3 days of dexamethasone therapy taken
7. Written informed consent from the patients or from close relatives of the patient if the patient is unconscious.

Exclusion Criteria:

1. History of anti-toxoplasmosis administrattion for more than 5 days before recruitment
2. Hypersensitivity or other contraindication to dexamethasone
3. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Mortality | 90 days
  Determined by the time from randomization to death (in days)

SECONDARY OUTCOMES:
Number of participants with grade 3 and 4 and serious adverse events related to study drug | 7 days
  Signs and symptoms of adverse event related to study drug including hypersensitivity, GI upset, respiratory, skin, musculoskeletal problems, vertigo, and electrolyte imbalance will be assessed daily for 7 days since the first administration of study drugs.
Changes in consciousness | 14 days
  Glasgow Coma Scale (GCS) will be used to quantify the level of consciousness. GCS is a continuous scale ranging from 3 - 15 with higher scores represent better outcome
  GCS will be recorded every day until day 14 of hospitalization
Neurological response (1) | up to 90 days
  Neurological responses that show both improvement (e.g. regaining consciousness) and worsening (i.e. decreasing of consciousness, development of new neurological deficits) will be measured and recorded at days 3, 7, 30, 60 and 90.
  Neurological response will be measured by serial assessments of Glasgow Outcome Scale (GOS).
  GOS is a scale that measures objective degree of recovery. It has 6 degrees of measurement ranging from 0 to 5, with 0 equals death and 5 full recovery.
Neurological response (2) | up to 90 days
  Neurological responses that show both improvement (e.g. regaining consciousness) and worsening (i.e. decreasing of consciousness, development of new neurological deficits) will be measured and recorded at days 3, 7, 30, 60 and 90.
  Second neurological response measurement will be using serial assessments of Modified Rankin Scale (mRS).
  The modified Rankin Scale (mRS) is commonly used for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0 to 6, with 0 equals to perfect health without symptoms, and 6 equals to death; i.e. the higher the score, the worse the outcome.
Cognitive function (1) | up to 90 days
  Cognitive function will be measured by using Mini Mental State Examination (MMSE) as early as the subjects regain consciousness and at day 7, 30 and 90.
  MMSE is a continuous scale with values from 0 to 30, and considered normal if the value is more than or equal to 28
Cognitive function (2) | up to 90 days
  The second cognitive function measurement will be using Montreal Cognitive Assessment Indonesian version (MoCA INA) as early as the subjects regain consciousness and at day 7, 30 and 90.
  MoCA-INA is a continuous scale with values from 0 to 30, and considered normal if the value is more than or equal to 26
Neuroradiological response | 90 days
  Change in brain oedema or development of any CT-scan abnormalities related to cerebral toxoplasmosis will documented by performing and comparing two series of CT-scan with contrast administration that will be done within the first 3 days and at day 90 (+/- 7 days) after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Sofiati Dian, M.D., PhD, Principal Investigator — Faculty of Medicine Universitas Padjadjaran Bandung
Locations (1):
- Hasan Sadikin General Hospital, Bandung, West Java, Indonesia